CLINICAL TRIAL: NCT06842186
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study of Ascending Doses of WVE-007 to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics in Adults Living With Overweight or Obesity
Brief Title: A Phase 1 Study of WVE-007 in Adults Living With Overweight or Obesity
Acronym: INLIGHT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wave Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WVE-007-001
Record Dates: First submitted 2025-01-29; First posted 2025-02-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-11

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Experimental): Experimental WVE-007 (Dose 1) or Placebo
  Interventions: Drug: WVE-007
- Cohort 2 (Experimental): Experimental WVE-007 (Dose 2) or Placebo
  Interventions: Drug: WVE-007
- Cohort 3 (Experimental): Experimental WVE-007 (Dose 3) or Placebo
  Interventions: Drug: WVE-007
- Cohort 4 (Experimental): Experimental WVE-007 (Dose 4) or Placebo
  Interventions: Drug: WVE-007
- Cohort 5 (Experimental): Experimental WVE-007 (Dose 5) or Placebo
  Interventions: Drug: WVE-007

INTERVENTIONS:
Drug: WVE-007 — Stereopure siRNA oligonucleotide

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of WVE-007 when administered subcutaneously (SC) as single ascending doses in adults who are affected by overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 18 to 60 years
* BMI 28 to 35 kg/m2 which has been stable (±5%) for the previous 3 to 6 months (based on participant self-report or medical records)
* Healthy, in the opinion of the Investigator, as determined by prestudy medical history, physical examination, and clinical laboratory assessments

Exclusion Criteria:

* History or presence of CV disease, including heart failure (New York Heart Association [NYHA] Class III or IV), myocardial infarction, angina, or clinically significant abnormal laboratory assessments
* History or presence of thyroid disorders
* Medical history or diagnosis of causes of liver disease
* Use of any siRNA agent in the prior 12 months
* Received an investigational agent within 90 days or 5 half-lives, whichever is longer, before the first dose of study drug or are in follow-up of another clinical study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with adverse events | Day 1 through end of study

SECONDARY OUTCOMES:
Maximum concentration of WVE-007 in plasma (Cmax) | Day 1 through 169
Area under the plasma concentration time curve for WVE-007 from time 0 to last measurable concentration (AUClast) | Day 1 through 169
Change over time from baseline levels of serum activin E | Day 1 through 169

OTHER OUTCOMES:
Percent change of weight (kg) from baseline | Day 1 through 169
Body composition changes as follows: Change in body fat percentage from baseline, percent change of visceral fat (kg) from baseline, and percent change in fat-free mass (kg) from baseline | Day 1 through 169

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Wave Life Sciences
Locations (6):
- Parexel International-EPCU Baltimore, Baltimore, Maryland, United States
- ARENSIA Research Clinic, Chisinau, Moldova
- Romania (2):
  - Arensia Clinics S.R.L., Bucharest
  - Spitalul Clinic Judetean De Urgenta Cluj, Cluj-Napoca
- United Kingdom (2):
  - Parexel International Early Phase Clinical Unit, Harrow
  - Simbec-Orion Clinical Pharmacology, Merthyr Tydfil

IPD SHARING:
Plan to Share IPD: No